CLINICAL TRIAL: NCT07274150
Title: Abdominal Aortic Junction Tourniquet (AAJT-S) for Non-compressible Torso Haemorrhage A Prospective Multicentre-study
Brief Title: Abdominal Aortic Junction Tourniquet (AAJT-S) for Non-compressible Torso Haemorrhage in the Prehospital and Emergency Room Setting
Status: Not yet recruiting | Type: Observational
Sponsor: Medical University of Graz (Other)
Responsible Party: Sponsor
Other Study IDs: 1331/2025
Record Dates: First submitted 2025-11-18; First posted 2025-12-10 (Actual); Last update posted 2025-12-10 (Actual); Status verified 2025-10

CONDITIONS: Exanguination; Polytrauma; NCTH
Keywords: NCTH; Exanguination; Aortic occlusion
MeSH Terms: conditions — Multiple Trauma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study seeks to evaluate the feasibility of a Abdominal Aortic Balloon Occlusion of the Aorta (AAJT-S) in exanguinating trauma patients with non-compressible truncal haemorrhage in the emergency room and the pre-hospital setting.

DETAILED DESCRIPTION:
Much like REBOA, AAJT-S can potentially stop blood flow distal to the device and therefore improve proximal aortic perfusion, minimize haemorrhage and stabilize patients until definite surgical repair/bleeding control is feasible. In contrast to REBOA, there is no need of femoral access and therefore, appropriate training is easily achieved.

This study seeks to gather further information on the benefits and potential harms of this intervention on a multicentre level.

ELIGIBILITY:
Inclusion Criteria:

1. Written consent of the participant after being informed
2. Aged, or believed to be aged, 18 years or above
3. Confirmed or suspected life-threatening lower body trauma (i.e. signs of inadequate perfusion of tissues, tachycardia, hypotension, suspected blood loss)
4. Thought to benefit from trauma resuscitation with AAJT-S or REBOA zone III
5. Traumatic cardiac arrest

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 1. Suspected additional bleeding source proximal to the umbilicus
  2. Known or suspected pregnancy at presentation
  3. Known abdominal aortic aneurysm
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2026-02-01 (Estimated); Primary Completion 2028-02-01 (Estimated); Study Completion 2028-07-01 (Estimated)

PRIMARY OUTCOMES:
effective placement of the device | 1 hour
  cessation of bloodflow distal to the device

SECONDARY OUTCOMES:
Outcome Measure | 30 days
  30-day in hospital mortality
Complications | 90 days
  Occurrence of complications of device application
hemodynamic improvement after application | 1 hour
  lower hart rate / higher blood pressure (improvement in bpm/mmHg)

CONTACTS AND LOCATIONS:
Locations (1):
- Medical University of Graz, Graz, Styria, Austria

IPD SHARING:
Plan to Share IPD: Undecided